CLINICAL TRIAL: NCT01578837
Title: Efficacy and Safety of Combined Rg3-enriched Korean Red Ginseng (Panax Ginseng C.A. Meyer) and American Ginseng (Panax Quinquefolius) as Poly-therapy in the Management of Concomitant Hypertension in Type 2 Diabetes
Brief Title: Combined Rg3-enriched Korean Red Ginseng and American Ginseng in the Management of Hypertension in Type 2 Diabetes
Acronym: R-KAT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OG-2-09-2920-VV
Record Dates: First submitted 2012-04-12; First posted 2012-04-17 (Estimated); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Diabetes Mellitus Type 2; Hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension | interventions — Asian ginseng; Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ginseng (Experimental): Combined Rg3-enriched Korean Red Ginseng and American Ginseng capsule
  Interventions: Dietary Supplement: Ginseng
- Wheat Bran (Placebo Comparator): 100 % Natural Wheat Bran capsule
  Interventions: Dietary Supplement: Wheat Bran

INTERVENTIONS:
Dietary Supplement: Ginseng — 2.25g of encapsulated ginseng (1.5g American Ginseng and 0.75g Rg3-enriched Korean Red Ginseng)will be administered in 6 identical capsules, 2 capsules with each meal (total 6 capsules per day).
  Arms: Ginseng
Dietary Supplement: Wheat Bran — 2.25g of encapsulated 100% natural wheat bran will be administered in 6 identical capsules, 2 capsules with each meal (total 6 capsules per day).
  Arms: Wheat Bran

SUMMARY:
The study is a combined Phase-I like (safety) and Phase-II like (efficacy) double blind randomized placebo controlled trial. The objective is to investigate whether the combination of AG and Rg3-enriched Korean Red ginseng added to conventional medical treatment are effective and safe in the long-term management of high blood pressure while managing type 2 diabetes. Eighty-five subjects with type 2 diabetes and concomitant high blood pressure (key inclusion criteria: HbA1c ≥ 6.5%- ≤ 8.0%) will be recruited for the study.

ELIGIBILITY:
Inclusion Criteria:

* between the age of 40 and 75 years
* type 2 diabetes (at least 1 year duration, HbA1c ≥ 6.5%- ≤ 8.0%, treated with diet and/or oral hypoglycemic medications)
* clinically diagnosed and treated hypertension according to Canadian Diabetes Association Clinical Practice Guidelines
* normal thyroid, kidney and liver functions
* female subjects recruited for the study must be post-menopausal or had absence of menstruation for ≥ 1 year or is taking contraceptive precautions

Exclusion Criteria:

* insulin therapy
* history of angina, myocardial infarction or stroke
* systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg
* use of ginseng within 1 month start of study
* BMI >35 kg/m2
* smoking cigarettes
* alcohol intake of > 2 drinks/day
* recently given blood
* have an upcoming planned surgery
* GFR <60 mL/min/1.73m2
* prolonged QT (>20 ms) interval as assessed by ECG
* changes to use of natural health products that may effect blood pressure and/or diabetes
* weight change more than +/- 3 kg/month
* HIV infection, inflammatory bowel disease, celiac disease, heart disease, bleeding disorder, sleep disorder, arrhythmia
* pregnant or breastfeeding
* use of anticoagulant (excluding aspirin), antiplatelet, sedative, sympathomimetic, photosensitizing or anti-depressant drugs
* hormone replacement therapy, furosemide, morphine, glucocorticoids
* presence of any conditions which, in the opinion of the Qualified Investigator, might jeopardize the health and safety of the subject or study personnel, or adversely affect the study results
* known sensitivity or allergy to any test product or placebo ingredients

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-04 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in Mean 24 hour Systolic Ambulatory Blood Pressure at 12 weeks | 12 Weeks

SECONDARY OUTCOMES:
Change in Mean 24 hour Diastolic, daytime and nighttime Ambulatory Blood pressure at 12 Weeks | 12 Weeks
Change in Pulse Pressure | 12 Weeks
Change in Central Augmentation Index and pulse wave analysis | 12 Weeks
Change in Pulse Wave Velocity at 12 Weeks | 12 Weeks
Change in low-grade body inflammation (hs-CRP) | 12 Weeks
Change in HbA1c | 12 Weeks
Change in Fasting Insulin | 12 Weeks
Change in Fasting Glucose | 12 Weeks
Change in Calculated HOMA-Insulin Sensitivity | 12 Weeks
Change in RHI at 12 weeks | 12 weeks
  vs control
Change in lipids at 12 weeks | 12 weeks
  vs control

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Vuksan, PhD, Principal Investigator — Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital
Locations (2):
- Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario, Canada
- Clinical Centre Vuk Vrhovac, Zagreb, Croatia

REFERENCES:
- [Derived] Jovanovski E, Smircic-Duvnjak L, Komishon A, Au-Yeung FR, Sievenpiper JL, Zurbau A, Jenkins AL, Sung MK, Josse R, Li D, Vuksan V. Effect of coadministration of enriched Korean Red Ginseng (Panax ginseng) and American ginseng (Panax quinquefolius L) on cardiometabolic outcomes in type-2 diabetes: A randomized controlled trial. J Ginseng Res. 2021 Sep;45(5):546-554. doi: 10.1016/j.jgr.2019.11.005. Epub 2019 Nov 14. PMID 34803424